CLINICAL TRIAL: NCT02385812
Title: Screening of Alberta Asbestos Exposed Workers for Lung Cancer and Mesothelioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment through COVID pandemic
Sponsor: University of Calgary (Other)
Collaborators: Alberta Cancer Foundation (Other); Western Canadian Mesothelioma Foundation (Unknown)
Responsible Party: Principal Investigator, Dr. Alain Tremblay, Professor, University of Calgary
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 10007822
Record Dates: First submitted 2014-11-27; First posted 2015-03-11 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer; Mesothelioma
Keywords: Lung Cancer; Mesothelioma; Asbestos; Screening
MeSH Terms: conditions — Lung Neoplasms; Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High lung cancer risk (Experimental): Individuals with lung cancer risk >= 1.5% over 6 years
  Interventions: Procedure: Low-dose computed tomography Annual scan x3
- Low lung cancer risk (Experimental): Individuals with lung cancer risk <1.5% over 6 years
  Interventions: Procedure: Low-dose computed tomography Baseline scan only

INTERVENTIONS:
Procedure: Low-dose computed tomography Annual scan x3 — Annual scan x3
  Arms: High lung cancer risk
Procedure: Low-dose computed tomography Baseline scan only — Baseline scan only
  Arms: Low lung cancer risk

SUMMARY:
Asbestos defines a group of naturally occurring mineral silicate fibers which are easily inhaled, resulting in a variety of diseases of the respiratory system including lung cancer and malignant mesothelioma. Despite some advances in treatment, there has been little impact on overall survival for both lung cancer and mesothelioma in the past 20 years in great part because patients usually present with disease at an advanced and incurable stage. This study aims to develop and implement a low-dose computed tomography (LDCT) screening approach for lung cancer and mesothelioma in asbestos-exposed workers in Alberta.

DETAILED DESCRIPTION:
In Canada, lung cancer is the primary cause of cancer mortality above the next three culprits combined (breast, colon and prostate cancer). Cigarette smoking is the most important risk factor in the development of lung cancer. Another population of particular interest in Alberta involves workers with occupational exposure to asbestos as asbestos and tobacco exposure results in a synergistic effect on lung cancer risk. Mesothelioma is a rare cancer of the lining of the lung with poor prognosis of which 80% of cases are believed to be related to asbestos exposure.

Unfortunately, despite some advances in treatment, there has been little impact on overall survival for both lung cancer and mesothelioma in the past 20 years in great part because patients usually present with disease at an advanced and incurable stage. Additional strategies are desperately needed to reduce the morbidity and mortality associated with this disease.

The objectives of this study are to develop and implement a LDCT screening approach for lung cancer and mesothelioma in asbestos-exposed workers in Alberta; to determine participants' motivation and expectations associated with a screening program, their satisfaction with the program, and the psychosocial consequences of the screening program; to determine the accuracy of a lung cancer risk prediction model modified to include asbestos exposure; and to determine the 3-year clinical incidence of lung cancer in asbestos-exposed individuals interested in lung cancer screening but who do not meet minimal risk threshold.

The investigators will offer a combined lung cancer and mesothelioma screening program for 200 Alberta asbestos-exposed workers based on low-dose CT scanning.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 - 80 years (either gender, any ethnic group)
* Documented exposure to asbestos for at least one year, at least 10 years prior to study entry
* Ability to provide informed consent and participate in study procedures

Exclusion Criteria:

* Any medical condition, such as severe heart disease (e.g. unstable angina, chronic congestive heart failure), severe lung disease or lung disease requiring supplemental oxygen, solid organ transplant, that in the opinion of the physician unlikely to benefit from screening due to shortened life-expectancy from the co-morbidities or inability to tolerate diagnosis and treatment of a screen detected abnormality
* Have been previously diagnosed with lung cancer or mesothelioma
* Have had other cancer within the past 5 years with the exception of the following cancers: non-melanomatous skin cancer, localized prostate cancer, carcinoma in situ (CIS) of the cervix, or superficial bladder cancer. Treatment of the exceptions must have ended >6 months before registration into this study
* Pregnancy
* CT scan of the chest in the past 2 years
* Unwilling to have a LDCT of chest
* Unwilling to sign a consent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01-01; Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in SF-12 quality of life score | Baseline vs. 14 days post receipt of screen results.

SECONDARY OUTCOMES:
Change in EQ-5D and STAI | Baseline vs. 14 days post receipt of screen results.
Lung cancer detection rate | 3 years
Mesothelioma detection rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alain Tremblay, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta